CLINICAL TRIAL: NCT07083167
Title: Anesthesia Clinical Practice During Labour Neuraxial Analgesia: A Prospective Observational Study
Brief Title: Anesthesia Clinical Practice During Labour Neuraxial Analgesia
Acronym: ACP-LNA
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Vit Gunka, Site Principal Investigator, University of British Columbia
Other Study IDs: H24-03381 ACP-LNA
Record Dates: First submitted 2025-06-13; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Labor Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anesthesiologists: All anesthesiologists providing labor neuraxial analgesia
  Interventions: Other: No Interventions.

INTERVENTIONS:
Other: No Interventions. — No interventions.

SUMMARY:
The goal of this observational study is to evaluate the communication between the anesthesiologist and the patient prior the initiation and during the administration of the labor neuraxial analgesia.

The investigators hypothesize that there will be differences among anesthesiologists during the informed consent process and communication during the procedure, specifically, how the anesthesiologists describe the technical aspects of the procedure, alternatives, risks, complications, and expected effects of labour neuraxial analgesia.

The anesthesiologists will be observed during a routine labor neuraxial analgesia procedure for healthy uncomplicated patients.

ELIGIBILITY:
Inclusion Criteria:

* all obstetric anesthesiologists working in maternity unit

Exclusion Criteria:

* any comorbidity of the patient that would necessitate deviation from a routine practice for the initiation of labor neuraxial analgesia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All obstetric anesthesiologists working in maternity unit
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Informed consent | From the first contact with the patient before labour neuraxial analgesia until the procedure is finished.
  Incidence of key elements (such as technique desciption, alternatives, risks, complications, and expected effects) during the consent process before the labour neuraxial analgesia procedure. This will be assessed using a structured observation checklist with dichotomous variables (yes/no).

SECONDARY OUTCOMES:
Procedure description | During the standard clinical consent process provided to patients prior to the administration of labour neuraxial anesthesia.
  Proportion of consent discussions in which the staff anesthesiologist described specific steps involved in administering labour neuraxial analgesia.
  Unit of measure: Percentage of specific consent discussions including each pre-defined procedural element using the data collection sheet (Appendix 3) during the observation of the consent process.
Additional labour analgesia options | During the standard clinical consent process provided to patients prior to the administration of labour neuraxial analgesia.
  Proportion of specific consent discussions in which the staff anesthesiologist offered additional labour analgesia options. Unit of measure: percentage of specific consent discussions in which alternative analgesia options were offered using the data collection sheet (Appendix 3) to document whether alternatives were discussed and which options (if any) were offered.
Risks and complications | During the standard clinical consent process provided to patients prior to the administration of labour neuraxial analgesia.
  Proportion of specific consent discussion in which specific risks and complications of labour neuraxial analgesia were mentioned and described to the patient in further detail. Unit of measure: percentage of specific consent discussions mentioning each risk; proportion thoroughly described versus briefly mentioned using the data collection sheet (Appendix 3).
Anticipated effects | During the standard clinical consent process provided to patients prior to the administration of labour neuraxial analgesia.
  Proportion of specific consent discussions that included discussion of what the patient should expect after the labour neuraxial anesthesia procedure. Unit of measure: percentage of specific consent discussions where each anticipated effect was mentioned (pre- and/or post-procedure) using the data collection sheet (Appendix 3).
Patient information sheets | During the standard clinical consent process provided to patients prior to the administration of labour neuraxial analgesia.
  Proportion of specific consent discussion in which the staff anesthesiologist being observed mentioned or offered the use of patient information sheets on labour neuraxial analgesia. Unit of measure: percentage of specific consent discussion involving the use or mention of an information sheet, which will be noted on the data collection sheet (Appendix 3) throughout the observed consent process.

CONTACTS AND LOCATIONS:
Overall Officials: Vit B Gunka, MD, Principal Investigator — Department of Anesthesia at BC Women's Hospital
Locations (1):
- Department of Anesthesia at BC Women's Hospital, University of British Columbia., Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yentis SM, Hartle AJ, Barker IR, Barker P, Bogod DG, Clutton-Brock TH, Ruck Keene A, Leifer S, Naughton A, Plunkett E. AAGBI: Consent for anaesthesia 2017: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2017 Jan;72(1):93-105. doi: 10.1111/anae.13762. PMID 27988961
- [Background] Tait AR, Teig MK, Voepel-Lewis T. Informed consent for anesthesia: a review of practice and strategies for optimizing the consent process. Can J Anaesth. 2014 Sep;61(9):832-42. doi: 10.1007/s12630-014-0188-8. Epub 2014 Jun 5. PMID 24898765
- [Background] Pattee C, Ballantyne M, Milne B. Epidural analgesia for labour and delivery: informed consent issues. Can J Anaesth. 1997 Sep;44(9):918-23. doi: 10.1007/BF03011961. PMID 9305553
- [Background] Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database Syst Rev. 2018 May 21;5(5):CD000331. doi: 10.1002/14651858.CD000331.pub4. PMID 29781504